CLINICAL TRIAL: NCT03119311
Title: A Novel Diagnostic Method for Exotropia Using Video-oculography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Sung-Hyuk Moon, professor, Inje University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IJ1234567
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Strabismus; Exotropia
MeSH Terms: conditions — Strabismus; Exotropia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOG group (Experimental): Video-oculography
  Interventions: Diagnostic Test: Video-oculography
- APCT group (Active Comparator): alternative prism cover test
  Interventions: Diagnostic Test: APCT

INTERVENTIONS:
Diagnostic Test: Video-oculography — Diagnostic Method for Exotropia Using Video-oculography
  Arms: VOG group
Diagnostic Test: APCT — alternative prism cover test
  Arms: APCT group

SUMMARY:
Thirty-four subjects with constant exotropia were included. Two independent ophthalmologists measured the angle of ocular deviation using alternate prism cover test (APCT). The video files and data with the changes in ocular deviation during the alternate cover test were obtained using video-oculography (VOG). To verify the accuracy of VOG, Investigator compared the value obtained using VOG and the angle of a rotating model eye, and subsequently made a new linear equation using these data. The calculated values obtained using VOG were compared with those obtained using APCT to determine the diagnostic accuracy of VOG.

ELIGIBILITY:
Inclusion Criteria:

* have horizontal strabismus, cooperative, visual acuity >= 1.0/1.0

Exclusion Criteria:

* have vertical strabimus> 5prism diopter, not cooperative, no agree

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
The angle of ocular deviation (degree,°) measured by VOG and PCT | 2 weeks after approval
  strabismic angle (degree,°) measured by VOG and PCT

CONTACTS AND LOCATIONS:
Locations (1):
- Busan Paik hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park N, Park B, Oh M, Moon S, Kim M. A quantitative analysis method for comitant exotropia using video-oculography with alternate cover. BMC Ophthalmol. 2018 Mar 22;18(1):80. doi: 10.1186/s12886-018-0747-9. PMID 29566654